CLINICAL TRIAL: NCT07268859
Title: Effect of Fan Application in Preventing Ticagrelor-associated Dyspnea in Patients With Acute Coronary Syndrome.
Brief Title: Effect of Fan Application in Preventing Ticagrelor-Associated Dyspnea
Acronym: ACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ATADEK2024-10/449; Is an identifier other (Other)
Record Dates: First submitted 2025-06-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Coronary Syndromes; Ticagrelor; Dyspnea
Keywords: Nursing; Ticagrelor; Hand fan therapy; Dyspnea; Non-pharmacological intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Dyspnea | interventions — CCP110 protein, human

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups: control and experimental. Randomization will be computer-based. Data will be analyzed by a statistician not involved in the study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by a statistician not involved in the study. Participants and researchers will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Control Group) (Active Comparator): Routine ward care including semi-Fowler position and breathing exercises. Standard institutional care will be applied. Presence, number, and severity of dyspnea attacks will be recorded during the first 2 hours after ticagrelor administration.
  Interventions: Other: STANDART CARE
- Standard Care + Fan Therapy (Experimental Group) (Experimental): In addition to standard care, patients will undergo hand fanning for 5 minutes at 30, 60, and 120 minutes after ticagrelor administration. The fan will be directed toward the patient's face from a distance of ~15 cm. Dyspnea severity and number of episodes will be recorded during this period.
  Device: Hand Fan
  Interventions: Other: STANDART CARE & FAN THERAPY

INTERVENTIONS:
Other: STANDART CARE — Routine ward care including semi-Fowler position and breathing exercises. Standard institutional care will be applied. Presence, number, and severity of dyspnea attacks will be recorded during the first 2 hours after ticagrelor administration.
  Arms: Standard Care (Control Group)
Other: STANDART CARE & FAN THERAPY — In addition to standard care, patients will undergo hand fanning for 5 minutes at 30, 60, and 120 minutes after ticagrelor administration. The fan will be directed toward the patient's face from a distance of ~15 cm. Dyspnea severity and number of episodes will be recorded during this period.
  Other Names: Fan
  Arms: Standard Care + Fan Therapy (Experimental Group)

SUMMARY:
This study will be conducted in the coronary intensive care unit of Dr. Siyami Ersek Chest, Heart and Vascular Surgery Training and Research Hospital. It aims to investigate the effect of hand fan therapy on ticagrelor-associated dyspnea in patients receiving ticagrelor.

DETAILED DESCRIPTION:
Patients in the coronary intensive care unit receiving ticagrelor and meeting the inclusion criteria will be included. The study includes two groups: a control group receiving standard care and an experimental group receiving standard care plus hand fan therapy. A total of 110 participants (55 per group) will be recruited. Randomization will be performed using a computer-based randomization program. Due to the nature of the intervention and sample characteristics, participants and the researcher will not be blinded. Data will be analyzed by a statistician not involved in the study, and the findings will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65,
* No severe hearing and vision problems,
* Can speak and understand Turkish,
* Easy to communicate with,
* First-time sufferer of acute coronary syndrome (ACS) for the first time,
* Decided to start ticagrelor therapy,
* Able to adapt to treatment,
* Individuals who volunteered to participate in the research.

Exclusion Criteria:

* Having any problem that prevents you from communicating cognitively, emotionally and verbally,
* Obstructive sleep abnormalities,
* Have a disease that affects respiratory function (stage IV cancer, bronchial asthma, COVID-19, lung cancer, pulmonary edema, chronic obstructive pulmonary disease, pulmonary hypertension, pulmonary embolism, pneumonia or bronchitis, etc.),
* With metabolic abnormalities,
* Intubated after the procedure,
* Previously treated with ticagrelor,
* Individuals who did not volunteer to participate in the study. Losses to follow up
* Individuals who wish to leave the study voluntarily.
* Saturation value below 95%,
* The one with the arrest,
* Who will not be able to fulfill the requirements of the work,
* Individuals with life-threatening conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of ticagrelor-associated dyspnea | Time Frame: 0-120 minutes after ticagrelor administration (T1: baseline; T2: 30 min; T3: 60 min; T4: 120 min) Unit of Measure: Percentage of participants (%)
  The proportion of participants who experience dyspnea within 120 minutes following ticagrelor administration will be recorded.

SECONDARY OUTCOMES:
Time to onset of ticagrelor-associated dyspnea | Time Frame: Within 120 minutes after ticagrelor administration (T1-T4) Unit of Measure: Minutes (min)
  The time interval between ticagrelor administration and the first reported dyspnea episode will be measured in minutes.

OTHER OUTCOMES:
Severity of ticagrelor-associated dyspnea | Time Frame: 0-120 minutes after ticagrelor administration (T1: baseline; T2: 30 min; T3: 60 min; T4: 120 min) Unit of Measure: Score (0-10)
  Dyspnea severity will be assessed using the Modified Borg Dyspnea Scale (0-10) at T1 (baseline), T2 (30 min), T3 (60 min), and T4 (120 min) after ticagrelor administration. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Üniversitesi-Cerrahapaşa, Istanbul, Avcılar
  - Sağlık Bilimleri Üniversitesi Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi Eğitim Araştırma Hastanesi, Istanbul, Üsküdar

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT07268859/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Ethics Approval (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT07268859/Prot_SAP_001.pdf
  • Informed Consent Form: Informed Consent Form (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT07268859/ICF_002.pdf